CLINICAL TRIAL: NCT05477082
Title: Use of Blood Gene Expression Profile and Donor-derived Cell-free DNA to Monitor Response to Treatment After Biopsy-proven Acute Rejection in Pediatric Kidney Transplant Recipients
Brief Title: Blood Biomarkers in Pediatric Kidney Transplant Recipients
Acronym: Omnigraf
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2022-30750
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Rejection of Kidney Allograft
Keywords: acute rejection; kidney transplant; pediatric; biomarker; cell free DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational group — Includes blood draws and data collection only

SUMMARY:
The objective of the proposed study is to assess whether a blood biomarker can be used to monitor the response to rejection treatment in pediatric kidney transplant recipients with biopsy-proven acute cellular or antibody mediated rejection. The study hypothesizes that blood gene expression profile and donor-derived cell-free DNA biomarkers (omnigraf) can be used to predict acute rejection and monitor its response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients
* Participants undergoing a for-cause kidney biopsy to rule out graft rejection
* Ages 21 years and less

Exclusion Criteria:

* Participants who have opted out of research
* Patients, less than 18 years of age, whose parents or legal guardians are illiterate and cannot read.
* Participants, 18 years and older, who are illiterate and cannot read.
* Participants, less than 18 years of age, whose parents or legal guardians do not speak English.
* Participants, 18 years and older, who do not speak English
* Participants who are pregnant as confirmed by medical records

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric kidney transplant recipients, ages < 21 years, scheduled to undergo a for-cause kidney biopsy to rule out graft rejection
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Biopsy-proven acute rejection | 7 days from baseline
  Yes or No assessment
Clinical resolution of rejection | 8 weeks from baseline
  Yes or No assessment; defined as improvement in serum creatinine to a value that is within 25% of baseline serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kizilbash, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States